CLINICAL TRIAL: NCT04926948
Title: SBRT With Immunotherapy for Mesothelioma
Brief Title: Stereotactic Body Radiation Therapy With Immunotherapy for the Treatment of Mesothelioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1924; NCI-2021-04302 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1924 (Other: Mayo Clinic in Rochester); 19-012226 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-05-21; First posted 2021-06-15 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Pleural Mesothelial Neoplasm
MeSH Terms: interventions — Immunotherapy; Adjuvants, Immunologic; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SBRT, immunotherapy) (Experimental): Patients undergo 3-5 daily fractions of SBRT in the absence of disease progression or unacceptable toxicity. Patients also receive immunotherapy at the discretion of the treating medical oncologist.
  Interventions: Other: Immunotherapy; Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Other: Immunotherapy — Immunotherapy
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial studies the effect of stereotactic body radiation therapy and immunotherapy in treating patients with mesothelioma. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving stereotactic body radiation therapy and immunotherapy may improve the tumors response to the treatment and decrease side-effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of focal stereotactic body radiation therapy (SBRT) with immune check inhibitors (ICI) for treatment of mesothelioma.

SECONDARY OBJECTIVES:

I. To determine progression free survival in patients treated with SBRT and ICI.

II. To assess acute and late toxicities overall in patients treated with SBRT and ICI.

TERTIARY OBJECTIVES:

I. To demonstrate that pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) levels correlate with tumor burden in patients with solid tumors.

II. To investigate if ctDNA can robustly identify molecular residual disease (MRD) before clinical, radiographic or pathologic progression in patients with solid tumors treated with definitive-intent surgery +/- radiotherapy +/- chemotherapy.

III. To determine whether post-resection ctDNA levels can be used to predict the risk of tumor recurrence and response to adjuvant radiation or adjuvant chemoradiation in patients with solid tumors.

IV. To determine if ctDNA levels can predict disease response and/or disease recurrence before clinical, pathologic or radiographic response/progression is confirmed in patients with solid tumors.

V. To perform methylation sequencing of cell-free DNA to noninvasively determine ctDNA cell- of-origin.

VI. To perform cell-free ribonucleic acid (RNA) analysis to monitor gene expression changes and identify genomic rearrangements.

VII. To perform epigenetic and genetic analyses including methylation sequencing and single cell RNA sequencing on associated tumor and peripheral blood cell samples.

EXPLORATORY OBJECTIVES:

I. To determine overall survival in these patients. II. To estimate the objective response rate (ORR) using immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST) 1.1 criteria.

III. To describe patterns of failure. IV. To estimate the quality of life (QOL) in these patients. V. Determine whether T-cell receptor expression changes during and after immunotherapy and SBRT, and whether these changes correlate with outcomes.

VI To evaluate potential predictive and prognostic biomarkers using various assays including flow cytometry assays, qualitative and quantitative analyses of patients' blood to explore associations with all primary and secondary endpoints.

OUTLINE:

Patients undergo 3-5 daily fractions of SBRT in the absence of disease progression or unacceptable toxicity. Patients also receive immunotherapy at the discretion of the treating medical oncologist.

After completion of study treatment, patients are followed up every 6 weeks for 36 weeks or per clinician discretion, then every 3 months for 2 years or until disease progression or study exit, then yearly for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of pleural mesothelioma
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Negative pregnancy test done =< 14 days prior to registration, for women of childbearing potential only. NOTE: male/female: Must be willing to use birth control for the entire study and must agree to use one of the following birth control methods listed:

  * Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
  * Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
  * Intrauterine device (IUD)
  * Abstinence (no sex)
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood samples for correlative research purposes
* Patient has received or is planning to receive ICI for mesothelioma
* Patient is planning to receive SBRT (stereotactic body radiation therapy) for mesothelioma

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treating patients with stereotactic body radiation therapy (SBRT) and immune checkpoint inhibitor | Up to 2 years
  Feasibility of treating patients with SBRT and ICI will be determined by ability to treat all enrolled patients without meeting stopping rules (maintaining <30%toxicity).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Defined as the time from study entry to any progression or death.
Incidence of acute toxicity | Up to 90 days post-SBRT
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will assess and summarize all acute and late AE's, regardless of attribution.
Incidence of late toxicity | Up to 90 days post-SBRT
  The maximum grade for each type of adverse event will be summarized using CTCAE version 5.0. Will assess and summarize all acute and late AE's, regardless of attribution.

OTHER OUTCOMES:
Response rate | Up to 2 years
  Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST). The frequency and percentage of responses will be calculated.
Patterns of failure | Up to 2 years
  Will be described descriptively as well using standard summary statistics (frequencies, percentages, etc.).
Quality of life (QOL) | Baseline up to 2 years
  Will be assessed using the Lung Cancer Symptom Scale (LCSS), which consists of nine questions assessing QOL in the past day. Questions are answered on a 10-point scale where 0=as good as it can be and 9=as bad as it can be. Lower score correspond to better QOL.
T-cell receptor expression changes | Baseline up to 2 years
  Will correlate changes with outcomes (PFS, OS, response, etc.). Potential predictive and prognostic biomarkers using various assays including flow cytometry assays, quality and quantitative analysis of patients' blood to explore associations with all primary and secondary endpoints will also be evaluated. Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the blood and tissue marker data will be correlated with clinical endpoints (PFS, OS, response, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, will use the Fisher's exact test. For biomarker data used to predict binary outcomes (i.e. response versus no response), will use logistic regression models.

CONTACTS AND LOCATIONS:
Overall Officials: William G. Breen, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials